CLINICAL TRIAL: NCT01707238
Title: Multi-Centre Clinical Evaluation Of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-39
Record Dates: First submitted 2012-09-21; First posted 2012-10-16 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stenfilcon A (Experimental): Participants wear a first pair of lenses for two weeks and then crossover and wear an alternate second pair of lenses for two weeks.
  Interventions: Device: etafilcon A
- etafilcon A (Active Comparator): Participants wear a first pair of lenses for two weeks and then crossover and wear an alternate second pair of lenses for two weeks.
  Interventions: Device: stenfilcon A

INTERVENTIONS:
Device: etafilcon A — Participants wear a first pair of lenses for two weeks and then crossover and wear an alternate second pair of lenses for two weeks.
  Other Names: etafilcon A (Daily Disposable Contact Lens)
  Arms: stenfilcon A
Device: stenfilcon A — Participants wear a first pair of lenses for two weeks and then crossover and wear an alternate second pair of lenses for two weeks.
  Other Names: stenfilcon A (Daily Disposable Contact Lens)
  Arms: etafilcon A

SUMMARY:
The purpose of this study is to compare the subjective performance for handling of two daily disposable contact lenses, stenfilcon A and etafilcon A.

DETAILED DESCRIPTION:
The study is to compare the subjective performance for handling of two daily disposable contact lenses, stenfilcon A and etafilcon A in this cross-over study.

ELIGIBILITY:
Inclusion Criteria:-

* Be between 16 and 45 years of age (inclusive)
* Adapted soft contact lens (CL) wearers (i.e. > 1 month)
* Spherical distance CL prescription between -1.00 and -6.00D (inclusive)
* Spectacle cylinder ≤0.75D in the least astigmatic eye, ≤1.00D in the other.
* Correctable to 6/9 (20/30) in both eyes
* Have the use of a mobile phone to send and receive text messages throughout the day for the duration of the study.
* Have read, understood and signed the informed consent
* Willing to comply with the wear schedule (at least 40 hours per week)
* Willing to comply with the study visit schedule

Exclusion Criteria:-

* Any active corneal infection, injury or inflammation
* Systemic or ocular allergies, which might interfere with CL wear
* Systemic disease, which might interfere with CL wear
* Ocular disease, which might interfere with CL wear
* Strabismus, amblyopia
* Subjects who have undergone corneal refractive surgery and any anterior segment surgery
* Subjects with keratoconus or other severe corneal irregularity contraindicating lens wear
* Pregnant or lactating
* Use of systemic/topical medication contraindicating CL wear
* Use of gas permeable contact lenses within the last month
* Employees of the investigational site or immediate family members of Investigators
* Participation in any concurrent clinical trial or in the last 30 days

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, Study Director — Visioncare Research Ltd.; Ruth Craven, Study Director — Visioncare Research Ltd.
Locations (7):
- United Kingdom (7):
  - Keith Tempany Opticians, Broadstone, Dorset
  - Cameron-Davies Optometrists, Southsea, Hampshire
  - Cameron-Davies Optometrists, Portchester, Hants
  - Leightons Opticians, St Albans, Hertfordshire
  - David Gould Opticians, Rawtenstall, Lancashire
  - Vision Express Optical Lab, Hendon, London
  - S.H. Harrold, Uxbridge, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number subjects enrolled per site ranged six to 25. Two sites were asked to enroll more than 20 subjects to fulfill required number of subjects. Approval from Ethics Committee sought before sites were invited to recruit additional subjects. Of the 100 enrolled, 13 were existing etafilcon A wearers, falling short of the 25% target.
Pre-assignment Details: All participants randomized to receive all interventions and combined into one Arm/Group, "Overall All Study Population" for the participant flow.
Groups:
- Stenfilcon A Then Etafilcon A: All subjects assigned as overall study population wore both sets of lenses. Overall study population was randomized to wear either stenfilcon A followed by etafilcon A or etafilcon A followed by stenfilcon A.
- Etafilcon A Then Stenfilcon A: All subjects assigned as overall study population wore both sets of lenses. Study population was randomized to wear either stenfilcon A followed by etafilcon A or etafilcon A followed by stenfilcon A.
Period: Overall Study
Arm/Group | Stenfilcon A Then Etafilcon A | Etafilcon A Then Stenfilcon A
Started | 48 | 52
Completed | 48 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects assigned as overall study population wore both sets of lenses. Study population was randomized to wear either stenfilcon A followed by etafilcon A or etafilcon A followed by stenfilcon A.
Groups:
- Etafilcon A Then Stenfilcon A: All subjects assigned as overall study population wore both sets of lenses. Overall study population was randomized to wear either stenfilcon A followed by etafilcon A or etafilcon A followed by stenfilcon A.
- Total: Total of all reporting groups
Arm/Group | Stenfilcon A Then Etafilcon A | Etafilcon A Then Stenfilcon A | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 11 | 17
  Between 18 and 65 years | 42 | 41 | 83
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 38 | 69
  Male | 17 | 14 | 31
Region of Enrollment [Number; unit: participants]
  United Kingdom | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Handling
Description: Participant's subjective rating for lens handling of Pair #1 surveyed at 2 weeks (+3) days after baseline visit and Pair #2 surveyed at 4 weeks (+3) days after baseline visit. Each pair worn for two weeks daily disposable wear basis (at least 40 hours per week). Lenses worn minimum 2 hours prior to visit. Rated by questionnaires (0-10, 10= very easy).
Time Frame: two weeks and four weeks from baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stenfilcon A; Etafilcon A: Participants randomized to wear a first pair of lenses for two weeks and then crossover and wear an alternate second pair of lenses for two weeks. (Stenfilcon A then etafilcon A and/or etafilcon A then stenfilcon A.)
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 100 | 100
units on a scale | 8.84 (1.56) | 6.76 (2.89)

2. Secondary Outcome: Comfort
Description: Participant's subjective rating for overall lens comfort of Pair #1 surveyed at 2 weeks (+3) days after baseline visit and Pair #2 surveyed at 4 weeks (+3) days after baseline visit. Lenses worn minimum 2 hours prior to visit. Rated by questionnaires (0-10, 10=can't feel).
Time Frame: two weeks and four weeks from baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 100 | 100
units on a scale | 8.84 (1.32) | 8.09 (1.83)

3. Secondary Outcome: Dryness
Description: Participant's subjective rating for overall lens dryness of Pair #1 surveyed at 2 weeks (+3) days after baseline visit and Pair #2 surveyed at 4 weeks (+3) days after baseline visit. Each pair worn for two weeks daily disposable wear basis (at least 40 hours per week). Lenses worn minimum 2 hours prior to visit. Rated by questionnaires (0-10, 10=no dryness).
Time Frame: two weeks and four weeks from baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 100 | 100
units on a scale | 8.51 (1.81) | 8.07 (1.50)

4. Primary Outcome: Satisfaction With Handling
Description: Participant's subjective rating for overall satisfaction of lens handling of Pair #1 surveyed at 2 weeks (+3) days after baseline visit and Pair #2 surveyed at 4 weeks (+3) days after baseline visit. Each pair worn for two weeks daily disposable wear basis (at least 40 hours per week). Lenses worn minimum 2 hours prior to visit. Rated by questionnaires (5 point Likert scale - Completely Dissatisfied, Somewhat Dissatisfied, Neither, Somewhat Satisfied, Completely Satisfied).
Time Frame: two weeks and four weeks from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 100 | 100
percentage of participants
  Completely Satisfied | 65 (0.85) | 28 (1.37)
  Somewhat Satisfied | 22 | 31
  Neither | 8 | 13
  Somwhat Dissatisfied | 5 | 16
  Completely Dissatisfied | 0 | 12

5. Secondary Outcome: Satisfaction With Dryness
Description: Participant's subjective rating for overall satisfaction of lens dryness of Pair #1 surveyed at 2 weeks (+3) days after baseline visit and Pair #2 surveyed at 4 weeks (+3) days after baseline visit. Each pair worn for two weeks daily disposable wear basis (at least 40 hours per week). Lenses worn minimum 2 hours prior to visit. Rated by questionnaires (5 point Likert scale - Completely Dissatisfied, Somewhat Dissatisfied, Neither, Somewhat Satisfied, Completely Satisfied).
Time Frame: two weeks and four weeks from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 100 | 100
percentage of participants
  Completely Satisfied | 58 (0.91) | 35 (1.00)
  Somewhat Satisfied | 30 | 43
  Neither | 5 | 8
  Somwhat Dissatisfied | 6 | 14
  Completely Dissatisfied | 1 | 0

6. Secondary Outcome: Satisfaction With Comfort
Description: Participant's subjective rating for overall satisfaction of lens comfort of Pair #1 surveyed at 2 weeks (+3) days after baseline visit and Pair #2 surveyed at 4 weeks (+3) days after baseline visit. Each pair worn for two weeks daily disposable wear basis (at least 40 hours per week). Lenses worn minimum 2 hours prior to visit. Rated by questionnaires (5 point Likert scale - Completely Dissatisfied, Somewhat Dissatisfied, Neither, Somewhat Satisfied, Completely Satisfied).
Time Frame: two weeks and four weeks from baseline visit
Measure: Number; unit: percentage of participants
Arm/Group | Stenfilcon A | Etafilcon A
Number analyzed (Participants) | 100 | 100
percentage of participants
  Completely Satisfied | 65 (0.82) | 51 (1.09)
  Somewhat Satisfied | 27 | 26
  Neither | 3 | 13
  Somwhat Dissatisfied | 4 | 7
  Completely Dissatisfied | 1 | 3

ADVERSE EVENTS:
Arm/Group | Stenfilcon A | Etafilcon A
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.